CLINICAL TRIAL: NCT03668873
Title: Telehealth Delivery of Treatment for Sleep Disturbances in Young Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cynthia Johnson, Director, Center for Autism; Professor, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AR170155
Record Dates: First submitted 2018-09-07; First posted 2018-09-13 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder; Sleep Disturbance
Keywords: Parent Training; Telehealth; Sleep Problems
MeSH Terms: conditions — Autism Spectrum Disorder; Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Parent Training (Experimental): The five SPT sessions (each 60-90 minutes in duration) are individually delivered over 10-week virtually (HIPAA compliant video-chat). After Session A, session order may be adjusted to address child-specific problems. One-on-one delivery of SPT permits flexibility for child-specific problems within the program.
  Interventions: Behavioral: Sleep Parent Training
- Sleep Parent Education (Active Comparator): SPE consists of five 60-90 minute sessions, delivered individually over 10 weeks. SPE provides useful information to families of young children with ASD and sleep problems. Session A is designed to develop rapport. The sleep hygiene session (Session B) has been modeled from the RUBI manual. The other sessions include a systematic presentation on several relevant topics. An example of a SPE session is provided in the Intervention section. This condition is intended to parallel what would be offered in typical care, but by telehealth, where a parent might be educated about ASD as well as attend an outpatient appointment at a sleep clinic.
  Interventions: Behavioral: Sleep Parent Education

INTERVENTIONS:
Behavioral: Sleep Parent Training — SPT provides a comprehensive intervention that teaches parents the basic concepts and practical skills to address an array of sleep problems.
  Arms: Sleep Parent Training
Behavioral: Sleep Parent Education — SPE is a structured program intended to mimic treatment as usual. Thus, SPE is an accepted treatment and serves as an active comparator that controls for time and attention.
  Arms: Sleep Parent Education

SUMMARY:
Study Design: Ninety children with Autism Spectrum Disorder (ASD), between the ages of 2 to less than 7 years, and their parents will be recruited for this 10 week randomized clinical trial. Participants will be randomized to five individually delivered sessions of Sleep Parent Training (SPT) or five individually delivered sessions of Sleep Parent Education (SPE). Delivery of the programs will be via telehealth platform which also includes parent-child coaching in real-time. In addition to baseline, outcome measures will be collected at week 5 (midpoint of trial) and week 10 (endpoint of trial) as well as follow-up at week 16 to determine durability of treatment.

DETAILED DESCRIPTION:
This study will deliver an already initially tested manualized parent training program specially targeting bedtime and sleep disturbances, but delivered via telehealth platform and enhancing the program using live parent coaching at bedtime. Utilizing REDCap automated survey invitations feature, investigators will provide reminders of the intervention recommendations and data collection requirements. In a randomized clinical trial of 90 children with ASD, ages 2 to less than 7 years, a parent training program targeting sleep disturbance (Sleep Parent Training; SPT), will be compared to Sleep Parent Education (SPE). The investigators hypothesize that SPT will be superior in improving child sleep, child daytime functioning as well as parent well-being compared to SPE.

Specific Aims: Aim 1. To evaluate the efficacy of Sleep Parent Training program (SPT) delivered via telehealth for sleep disturbances compared Sleep Parent Educational Program (SPE, time and attention control) also delivered via telehealth in 90 children with ASD (ages >2 to <7 years) with moderate or greater sleep disturbances as measured by the Composite Sleep Index (CSI) of the modified Simonds and Parraga Sleep Questionnaire (MSPSQ).97 Aim 2. To evaluate the impact of SPT on child and parent quality of life (daytime child behavior, parental stress, parent sense of competency, mental health) compared to SPE.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders >2 and <7 years of age
2. Clinical diagnosis of ASD corroborated by the Modified Checklist for Autism in Toddlers169 or the Social Communication Questionnaire.170
3. Score of >5 on the CSI and a Clinical Global Impression Severity (CGI-S) score of Moderate or greater.
4. Medication and supplement free or on stable medication or supplements (no changes in the past 6 weeks and no planned changes for 16 weeks).
5. Parental proficiency in spoken and written English language.

Exclusion Criteria:

1. Children with a serious medical condition or a known or suspected medical cause for sleep disturbances (e.g., nocturnal seizures, unresolved gastrointestinal problems such as reflux or constipation).
2. Children with a psychiatric disorder or serious behavioral problems requiring immediate treatment.
3. Children with known or suspected sleep apnea, restless legs, or periodic limb movements during sleep, or a circadian-based sleep disorder (e.g. delayed or advanced sleep phase syndrome) based on history and all available information.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Johnson, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Centerl for Autism, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Shared in NDA

REFERENCES:
- [Result] Johnson CR, Turner KS, Foldes E, Brooks MM, Kronk R, Wiggs L. Behavioral parent training to address sleep disturbances in young children with autism spectrum disorder: a pilot trial. Sleep Med. 2013 Oct;14(10):995-1004. doi: 10.1016/j.sleep.2013.05.013. Epub 2013 Aug 27. PMID 23993773
- [Result] Johnson CR, Barto L, Worley S, Rothstein R, Alder ML. Telehealth parent training for sleep disturbances in young children with autism spectrum disorder: A randomized controlled trial. Sleep Med. 2023 Nov;111:208-219. doi: 10.1016/j.sleep.2023.08.033. Epub 2023 Sep 12. PMID 37806263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in November 2018 and the final participant was enrolled in August 2022.
Pre-assignment Details: 140 children were pre-screened and 102 were found to be eligible for a full screen. Of those, 91 consented. There were 14 screen failures (4 whose CSI was less than 5, 7 whose ASD diagnosis could not be corroborated, and 3 who did not follow through with full screening). Leaving 77 participants to be randomized, data were available for 36 participants randomized to SPT and 38 participants to SPE after 2 drop out in SPT and 1 in SPE before the intervention was initiated.
Groups:
- Sleep Parent Training: The five SPT sessions (each 60-90 minutes in duration) are individually delivered over 10-weeks. In addition to the five sessions, there are three home visits conducted via Express Care Online (HIPAA compliant video-chat). After Session A, session order may be adjusted to address child-specific problems. One-on-one delivery of SPT permits flexibility for child-specific problems within the program.
  Sleep Parent Training: SPT provides a comprehensive intervention that teaches parents the basic concepts and practical skills to address an array of sleep problems.
- Sleep Parent Education: SPE consists of five 60-90 minute sessions, delivered individually over 10 weeks. SPE provides useful information to families of young children with ASD and sleep problems. Session A is designed to develop rapport. The sleep hygiene session (Session B) has been modeled from the RUBI manual. The other sessions include a systematic presentation on several relevant topics. An example of a SPE session is provided in the Intervention section. This condition is intended to parallel what would be offered in typical care, but by telehealth, where a parent might be educated about ASD as well as attend an outpatient appointment at a sleep clinic.
  Sleep Parent Education: SPE is a structured program intended to mimic competent treatment as usual. Thus, SPE is an accepted treatment and serves as an active comparator that controls for time and attention.
Period: Overall Study
Arm/Group | Sleep Parent Training | Sleep Parent Education
Started | 38 | 39
Completed | 32 | 36
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Parent Training | Sleep Parent Education | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.6 (1.4) | 3.8 (1.4) | 3.7 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 29 | 33 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 29 | 24 | 53
  More than one race | 2 | 7 | 9
  Unknown or Not Reported | 0 | 1 | 1
Type of group educational activity the child attends, n (%)* [Count of Participants; unit: Participants]
  Child Care only | 2 | 4 | 6
  Public School | 7 | 7 | 14
  Private School | 5 | 3 | 8
  Special Education | 13 | 14 | 27
  None | 9 | 9 | 18
  Data Missing | 0 | 1 | 1
Child's usual living arrangement, n (%) [Count of Participants; unit: Participants]
  Parental Home (At Least One Parent) | 35 | 37 | 72
  Relative (Other Than Parents) | 1 | 1 | 2
In the current household, primary caregiver's highest level of education, n (%) [Count of Participants; unit: Participants]
  High school graduate or GED | 4 | 4 | 8
  Some college or post-high school or 2yr degree | 5 | 4 | 9
  College Graduate | 13 | 9 | 22
  Advanced graduate or professional degree | 14 | 21 | 35
Modified Simonds & Parraga Sleep Questionnaire-Composite Sleep Index (baseline), mean ± sd [Mean (Standard Deviation); unit: units on a scale] — The CSI was calculated by assigning a score to bedtime resistance item 5, night waking item 10, early waking item 51 and sleeping in places other than bed item 35. Scores were assigned for the duration of sleep latency item 6 and night wakings item 12. The total CSI score ranged from 0 to 12 with higher scores indicating more severe bedtime and sleep patterns. Minimum score of 5 required for participation. A change of 2 points or more is clinically significant.
  units on a scale | 7.6 (2.2) | 7.4 (2.0) | 7.5 (2.1)
Clinical Global Impressions - Severity (baseline), mean ± sd [Mean (Standard Deviation); unit: units on a scale] — This 7-point scale ranges from 1 (Normal) through 4 (Moderate) to 7 (Extreme) is a measure of severity of the child's condition. Although sleep problems will be given particular weight, the independent evaluator (IE) consider all aspects of the child's functioning to assign the CGIS score.
  units on a scale | 3.9 (.65) | 4 (.75) | 4 (0.70)
Aberrant Behavior Checklist Subscale I (Irritability) (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — Each item is rated on a Likert scale from 0 (not a problem) to 3 (severe in degree). The 15 item Irritability subscale has a range from 0- 45, higher score indicating more severity.
  units on a scale | 16 (10) | 13 (7.8) | 14 (9.2)
Aberrant Behavior Checklist Subscale II (Social Withdraw) (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — ABC Scale- each item is rated on a Likert scale from 0 (not a problem) to 3 (severe in degree). Subscale II (Social withdrawal)- 16 items range from 0- 48, higher score indicating more severity.
  units on a scale | 14 (8.5) | 11 (6.9) | 13 (7.9)
Aberrant Behavior Checklist Subscale III (Stereotypic Behavior) (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — ABC Scale- each item is rated on a Likert scale from 0 (not a problem) to 3 (severe in degree). Subscale III (Stereotypic behavior)- 7 items, range 0 to 21, higher score indicating more severity.
  units on a scale | 7 (5.1) | 5.5 (5.1) | 6.2 (5.1)
Aberrant Behavior Checklist Subscale IV (Hyperactivity/Noncompliance) (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — Each item is rated on a Likert scale from 0 (not a problem) to 3 (severe in degree). Hyperactivity subscale has 16 items, range 0- 48, higher score indicating more severity.
  units on a scale | 25 (12) | 22 (12) | 23 (12)
Aberrant Behavior Checklist Subscale V (Inappropriate Speech) (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — Each item is rated on a Likert scale from 0 (not a problem) to 3 (severe in degree). Inappropriate speech subscale has 4 items, range 0- 12, higher score indicating more severity.
  units on a scale | 3.1 (2.8) | 3 (2.6) | 3.1 (2.7)
Children's ChronoType Questionnaire Morningness/Eveningness (M/E) scale score (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — M/E scale-scores range from 10 (extreme morningness) to 49 (extreme eveningness). Morning types are classified by a M/E scale score of ≤23, intermediate types by a score of 24-32, and evening types by a score ≥33.
  units on a scale | 26 (7.1) | 28 (8.4) | 27 (7.8)
Parenting stress index-short form Defensive Responding (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — The Parenting Stress Index- Short Form(PSI) is rated on a 5-point scale (from "Strongly Disagree" = 1 to "Strongly Agree" = 5). Defensive Responding is ranged from 7- 35. Significant is less than 10.
  units on a scale | 21 (5.9) | 20 (7.4) | 21 (6.7)
Parental Stress Index Parental Distress (PD) (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — The Parenting Stress Index- Short Form(PSI) is rated on a 5-point scale (from "Strongly Disagree" = 1 to "Strongly Agree" = 5). PD scale range is 12-60, higher score is more severe.
  units on a scale | 33 (8.9) | 33 (11) | 33 (10)
Parental Stress Index Parent-Child Dysfunctional interaction (P-CDI) (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — The Parenting Stress Index- Short Form(PSI) is rated on a 5-point scale (from "Strongly Disagree" = 1 to "Strongly Agree" = 5). P-CDI scale range is 12-60, higher score is more severe.
  units on a scale | 34 (7.1) | 32 (6.6) | 33 (6.9)
Parental Stress Index Difficult Child (DC) (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — The Parenting Stress Index- Short Form(PSI) is rated on a 5-point scale (from "Strongly Disagree" = 1 to "Strongly Agree" = 5). DC scale range is 12-60, higher score is more severe.
  units on a scale | 43 (6.2) | 40 (6.5) | 41 (6.4)
Parenting stress index-short form- Total Stress (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — Parenting Stress Index- Short Form (PSI) is a 36-item parent questionnaire rated on a 5-point scale (from "Strongly Disagree" = 1 to "Strongly Agree" = 5). The PSI total stress ranges from 36 to 180, higher score being more stressed. A total score of 88 (85th percentile) and above is considered in the clinically significant range for parental stress.
  units on a scale | 111 (16) | 105 (21) | 108 (19)
Parenting Sense of Competence Scale Total Score (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — The Parenting Sense of Competence (PSOC) is a 17-item rating scale that assesses parental feelings of satisfaction and efficacy as a parent. Rated on a 6-point scale (from "Strongly Agree" = 1 to "Strongly Disagree" = 6.) Range 17- 102. The PSOC also yields a Total Competence score, with higher scores reflecting higher competence.
  units on a scale | 72 (11) | 72 (14) | 72 (13)
Patient Health Questionnaire Total Score (baseline), mean ± sd* [Mean (Standard Deviation); unit: units on a scale] — 3-point scale (from "Not at all" = 0 to "Nearly everyday" = 3). Higher score shows more severity. Range 0 to 12.
  units on a scale | 4 (2.7) | 4 (3.5) | 4 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on MSPSQ-CSI
Description: Modified Simonds & Parraga Sleep Questionnaire-Composite Sleep Index (MSPSQ - CSI). The modified version of the Simonds & Parraga Sleep Questionnaire (MSPSQ6 was completed by the child's primary caregiver at baseline, and weeks 5 and 10 weeks for both groups. We used earlier described conventions for determining the MSPSQ - CSI score. The CSI was calculated by assigning a score to the frequency of sleep problems targeted: bedtime resistance (item 5), night waking (item 10), early waking (item 51) and sleeping in places other than bed (item 35). In addition, scores were assigned for the duration of sleep latency (item 6) and night wakings (item 12). Minimum score of 0 and maximum score of 12, higher score indicated worse outcome. The sample sizes reflect the number of participants who completed surveys at each follow-up.
Time Frame: Baseline, 5 weeks, and 10 weeks
Population: A modified intention-to-treat principle was used for the primary analysis, in which participants who attended at least one treatment session were analyzed in the group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sleep Parent Training | Sleep Parent Education
Number analyzed (Participants) | 32 | 33
units on a scale
  Week 5 | -2.09 [-3.05 to -1.12] | -0.64 [-1.24 to -0.04]
  Week 10: number analyzed (Participants) | 32 | 32
  Week 10 | -3.31 [-4.08 to -2.54] | -1.46 [-2.19 to -0.73]
Statistical Analysis 1: Comparison: Sleep Parent Training vs Sleep Parent Education; The null hypothesis was that the SPE and SPT groups did not differ on change in CSI score at 10 weeks. Assuming a standard deviation of 2.5 units and an attrition rate of 10%, an enrollment target of 90 participants would provide 90% power to detect a difference of 1.85 points or greater with a type I error rate of 0.05 using a two-tailed two-sample t-test; Test type: Superiority; p < 0.001, Mixed Models Analysis — Threshold for significance was p=0.05; Mixed models with repeated measures with fixed effects for baseline CSI, treatment, week as a categorical variable, and treatment-week interaction; Difference of Least Squares Means = -1.85, 95% CI 2-sided [-2.88 to -0.81] — Treatment difference = SPT minus SPE

2. Primary Outcome: Percentage of Treatment Responders at Week 10 Using Clinical Global Impression (CGI-I) Scale
Description: Improvement scale of the Clinical Global Impression (CGI-I) Scale is a clinician-rated, 7-point scale designed to measure overall improvement from baseline. Scores range from 1 (Very Much Improved) to 4 (Unchanged) to 7 (Very Much Worse). An IE masked to group assignment used all available information to judge treatment response. CGI-I ratings of Much Improved (score of 2) or Very Much Improved (score of 1) were used to classify subjects as positive responders. All other scores classify subjects as negative responders. Subjects who dropped out or had missing data were classified as negative responders.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Parent Training | Sleep Parent Education
Number analyzed (Participants) | 36 | 38
Participants | 20 | 12
Statistical Analysis 1: Comparison: Sleep Parent Training vs Sleep Parent Education; The null hypothesis was that the SPE and SPT groups did not differ on the rate of positive response to CGI-I at 10 weeks. Assuming a 25%-40% positive response rate at 10 weeks in the SPE group and 45 patients per group, power was 90% to detect a 32% or greater difference in positive response rate (57%-72% in SPT group, respectively), with a type I error rate of 0.05 using a Chi-square test; Test type: Superiority; p = 0.037, Chi-squared — Threshold for significance was 0.05; Absolute percent difference = 24, 95% CI 2-sided [2 to 46] — Difference = SPT minus SPE

3. Secondary Outcome: Change in ABC- Irritability From Baseline
Description: Aberrant Behavior Checklist. Each item is rated on a Likert scale from 0 (not a problem) to 3 (severe in degree)The ABC has shown adequate sensitivity to change in several pharmacological and behavioral treatment studies. The 15 item Irritability subscale has been used in other studies as a proxy for sleep-related impairment. Scores range from 0 to 45, higher score meaning a worse outcome. The sample sizes reflect the number of participants who completed surveys at each follow-up
Time Frame: Baseline, 5 weeks, and 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sleep Parent Training | Sleep Parent Education
Number analyzed (Participants) | 31 | 33
units on a scale
  week 5 | -0.13 [-2.28 to 2.01] | -2.00 [-3.29 to -0.70]
  week 10: number analyzed (Participants) | 31 | 32
  week 10 | -2.32 [-4.29 to -0.36] | -2.6 [-3.78 to -1.43]
Statistical Analysis 1: Comparison: Sleep Parent Training vs Sleep Parent Education; Test type: Superiority; p = 0.81, Mixed Models Analysis — threshold for significant 0.05

4. Secondary Outcome: Change in PSI From Baseline
Description: This 36-item parent-completed questionnaire for children 12 years of age and younger and has three scales: 1) Parental Distress; 2) Difficult Child Characteristics; and, 3) Dysfunctional Parent-Child Interaction. This measure was developed from the PSI Full Form using factor analysis, and has been used to assess parental stress and parent-child relationships in children with autism and intellectual disabilities. Scores range from 36- 180. A total score of 88 (85th percentile) and above is considered in the clinically significant range for parental stress. The sample sizes reflect the number of participants who completed surveys at each follow-up
Time Frame: baseline, 5 weeks, and 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sleep Parent Training | Sleep Parent Education
Number analyzed (Participants) | 30 | 33
units on a scale
  Week 5 | -6.23 [-10.38 to -2.07] | -4.94 [-9.88 to 0.00]
  Week 10: number analyzed (Participants) | 30 | 32
  Week 10 | -9.88 [-15.05 to -4.72] | -8.77 [-14.22 to -3.33]
Statistical Analysis 1: Comparison: Sleep Parent Training vs Sleep Parent Education; Test type: Superiority; p = 0.77, Mixed Models Analysis — Threshold for significance was 0.05

5. Secondary Outcome: PSOC Change From Baseline
Description: This 17-item scale was developed to assess parental self-efficacy. Each item is answered on a 6-point scale ranging from strongly disagree to strongly agree. The PSOC also yields a Total Competence score ranging from 17 to 102 with higher scores reflecting higher competence.
Time Frame: Baseline, 5 week, 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sleep Parent Training | Sleep Parent Education
Number analyzed (Participants) | 31 | 32
units on a scale
  Week 5 | 2.9 [0.81 to 4.99] | -1.81 [-4.41 to 0.78]
  Week 10 | 3.96 [1.98 to 5.94] | -0.68 [-3.04 to 1.68]
Statistical Analysis 1: Comparison: Sleep Parent Training vs Sleep Parent Education; Test type: Superiority; p = 0.003, Mixed Models Analysis — Threshold for significance was 0.05

6. Other Pre Specified Outcome: Treatment Fidelity
Description: Treatment fidelity checklists include the therapist integrity goals, parent objectives and level of adherence for each SPT and SPE session. Therapists rate themselves on 5-7 session-specific goals on a scale of 0 to 2 as follows: (0 = Goal was not achieved; 1 = Goal was partially achieved; 2 = Goal was fully achieved). Therapists are asked to comment on items rated 0. Parent objectives and adherence are scored on a similar scale. The score for each session = sum of scores for all items in that session divided by the total possible score X 100 (possible range 0-100%, higher score is better fidelity and adherence). The treatment fidelity checklists have been modeled after four other previously NIH-funded projects.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage
Arm/Group | Sleep Parent Training | Sleep Parent Education
Number analyzed (Participants) | 36 | 38
percentage
  Treatment Integrity | 98.05 [40 to 100] | 98.27 [66.6 to 100]
  Parent Adherence | 97.69 [60 to 100] | 99.15 [50 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at screening, baseline, week 5, week 10 and week 16.
Description: The Safety/Adverse Event Review Form also asked about the child's sleep, appetite and bowel habits. Reports of new adverse events or worsening of previously reported events were rated mild, moderate or severe. Hospitalization was documented as a serious adverse event. A "yes" answer to any of these queries prompted further questions to determine duration and severity. The onset, offset and severity of adverse events was documented whether presumed to be related to the study treatment or not.
Arm/Group | Sleep Parent Training | Sleep Parent Education
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/36
Other Adverse Events (participants affected / at risk) | 15/32 | 14/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sleep Parent Training (N=32) | Sleep Parent Education (N=36)
PICA event (Gastrointestinal disorders) | 1 (1) | 1 (1) — Eating of non-food items that resulted in emergency department visitation for observation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sleep Parent Training (N=32) | Sleep Parent Education (N=36)
cold or unknown virus (Infections and infestations) | 9 | 11 — cold or unknown virus
Tooth injury (General disorders) | 2 | 1 — Chipped tooth or lost tooth
COVID-19 (Infections and infestations) | 1 | 0 — COVID-19 Positive
Constipation (General disorders) | 2 | 1
Ear Infection (Infections and infestations) | 1 | 2

LIMITATIONS AND CAVEATS:
In designing the trial for telehealth delivery, we did not include some measures we might have if the study was in-person. For example, we did not have cognitive or language measures. These could also be treatment moderators in a larger study. We also did not include a measure of anxiety which is a likely predictive for treatment response. Further absent were measures of repetitive / restrictive behaviors or sensory sensitivities; both domains may influence response to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT03668873/Prot_SAP_000.pdf